CLINICAL TRIAL: NCT02164695
Title: Cardioprotective Effects of Remote Ischemic Perconditioning in Patients With ST-segment Elevation Myocardial Infarction Treated With Primary Percutaneous Coronary Intervention
Brief Title: Remote Ischemic Perconditioning in Patients With ST-segment Elevation Myocardial Infarction
Acronym: CAPRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Young Jin Youn, MD, PhD, Professor, Division of Cardiology, Department of Internal Medicine, Yonsei Univeristy Wonju College of Medicine, Yonsei University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR314003
Record Dates: First submitted 2014-06-12; First posted 2014-06-16 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: ST-segment Elevation Myocardial Infarction
Keywords: ST-segment elevation myocardial infarction; Remote ischemic perconditioning; Primary percutaneous coronary intervention; Cardiac magnetic resonance
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: * Control group: PPCI only
  * Study group: PPCI + RIPC
Who Masked: Outcomes Assessor
Masking Description: CMR results will be interpreted by observers blinded to randomization
Oversight: Data Monitoring Committee: No

ARMS (2):
- PPCI plus RIPC (Active Comparator): The patients randomized to PPCI plus RIPC group will receive RIPC during PPCI.
  Interventions: Procedure: PPCI plus RIPC
- PPCI only (Sham Comparator): The patients randomized to PPCI only group will receive PPCI only but the sham procedure of RIPC.
  Interventions: Procedure: PPCI only

INTERVENTIONS:
Procedure: PPCI plus RIPC — All patients will be prepared with an upper-arm blood pressure cuff before arterial puncture (contralateral in case of radial access). In patients allocated into PPCI plus RIPC group, the protocol will be started immediately after cuff preparation. Upper-arm will be exposed to 4 cycles of ischemia/reperfusion, each obtained by 5 min cuff inflation at 200mmHg, followed by 5 min complete deflation.
  Arms: PPCI plus RIPC
Procedure: PPCI only — All patients randomized to PPCI only arm, the blood pressure cuff will be applied to the arm or the calf but will not be inflated.
  Arms: PPCI only

SUMMARY:
To evaluate whether remote ischemic per-conditioning (RIPC) can reduce infarct size in patients with ST-segment elevation myocardial infarction treated with primary percutaneous coronary intervention (PPCI) within 12 hours of symptoms onset.

* Control group: PPCI only
* Study group: PPCI + RIPC

Primary endpoint: Infarct size measured by contrast-enhanced cardiac magnetic resonance (CMR) at 6 months after the index procedure

DETAILED DESCRIPTION:
ST-elevation myocardial infarction (STEMI) is a leading cause of mortality and morbidity. Early myocardial reperfusion with either of thrombolytic therapy or primary percutaneous coronary intervention (PPCI) is the most effective strategy for reducing the size of a myocardial infarct and improving the clinical outcome. Although this process can restore blood flow to the ischemic myocardium, it can induce injury. This phenomenon termed myocardial reperfusion injury can paradoxically reduce the beneficial effects of myocardial reperfusion. The pre-clinical study in animal models of acute myocardial infarction suggests that lethal reperfusion injury accounts for up to 50% of the final size of a myocardial infarct.

Remote ischemic conditioning uses brief ischemia and reperfusion of a distant organ to protect the myocardium. In animal study, remote ischemic postconditioning seems to be more effective than local postconditioning in experimental myocardial infarction.Bøtker et al. has reported remote ischemic preconditioning before hospital admission increase myocardial salvage in patients with acute myocardial infarction.

The objective of this study is to evaluate whether remote ischemic per-conditioning (RIPC) can reduce late infarct size in patients with STEMI treated with PPCI within 12 hours of symptoms onset. To test this hypothesis, we will randomize patients into PPCI + RIPC or PPCI alone. We will evaluate marker of reperfusion injury using contrast cardiac magnetic resonance image.

ELIGIBILITY:
Inclusion Criteria:

* Age >19 years
* Presenting within 12 hours of symptom onset
* >20 min of chest pain
* ST-elevation myocardial infarction defined as ST-segment elevation (>0.1 mV) in at least 2 contiguous precordial leads

Exclusion Criteria:

* Previous myocardial infarction
* Presence of chronic total occlusion
* Evidence of retrograde filling by collaterals at coronary angiography (Rentrop 2 or 3 collateral flow)
* Severe multi-vessel coronary artery disease to require further interventions before follow-up CMR
* Cardiac arrest before randomization
* Arrhythmias requiring external electric shock before randomization
* Unwillingness to participate
* External electric shock for cardioversion within first 3 days
* Cardiac surgery within first 3 days

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Infarct size measured by contrast-enhanced cardiac magnetic resonance | 6 months after index procedure
  Infarct size will be assessed on late-contrast images (≈10 min after gadolinium administration) by manually tracing the hyperintense area in each short-axis slice.

SECONDARY OUTCOMES:
Enzymatic Infarct Size | 1 to 5 days after index procedure
  Enzymatic infarct size will be assessed by the area under the curve of creatine kinase-myocardial band (CK-MB) and troponin I (TnI) release. Blood samples will be collected before PCI and every day after index PPCI. Area under the curve of CK-MB and troponin I release will be expressed in arbitrary units and calculated with the trapezoidal method.
Resolution of ST-segment deviation | 1 to 5 days after index procedure
  ST-segment deviation score will be measured in 12-lead electrocardiograms, calculated as the sum (in millimeters) of ST-segment deviation (elevation or depression) at 80 ms after the J-point in all 12 leads. ST-segment deviation score will be measured at presentation and 30 min after PCI, by 2 physicians blinded as to the patients' data, and the mean value of the 2 assessments will be used. ST-segment resolution will be calculated as a percentage: ratio of the reduction in ST-segment deviation score from presentation to half an hour after PCI over the ST-segment deviation score at presentation × 100% (i.e., [(ST-segment deviation at presentation - ST-segment deviation post-PCI)/ST-segment deviation at presentation] × 100%). Full ST-segment resolution will be defined as 80% or more reduction of ST-segment deviation score.
Acute kidney injury | 1 to 3 days after index procedure
  Acute kidney injury will be defined as an absolute increase in serum creatinine of ≥0.5 mg/dl or a relative increase of ≥25% compared with baseline within 96 h after PCI (the maximal measured concentration of serum creatinine during these 96 h will be used). Relative reduction in estimated glomerular filtration rate (eGFR), calculated with the Modification of Diet in Renal Disease formula, within 96 h after PCI will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Young Jin Youn, MD, Principal Investigator — Yonsei Univeristy Wonju College of Medicine
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea